CLINICAL TRIAL: NCT04450420
Title: Tunnel Construction Course Pilot Assessment of Simulation-based Training Effectiveness
Acronym: TCC-PASTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HelpMeSee Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TCCPASTE
Record Dates: First submitted 2020-06-19; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Cataract
Keywords: cataract; MSICS; manual small incision cataract surgery; surgical simulation; simulation
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Expert raters assessing outcomes by watching videos of surgery were masked to the identity of the participating surgeon, their institutional affiliation, and the sequence in which they performed procedures in the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation based curriculum (Experimental): Three phases:
  1. Self-study of an eBook - Participating trainees will be required to learn material pertaining to tunnel construction and general surgical principles during SICS from an eBook that has been developed by HelpMeSee.
  2. Instructor led teaching - didactic training, lab activities to gain familiarity with instruments, simulator based training through deliberate practice, and debriefing with instructor.
  3. Instructor supervised performance of surgery on patients in the operating room.
  Interventions: Other: Simulation based curriculum
- Standard training (Active Comparator): Current standard curriculum for resident training.
  Interventions: Other: Standard training

INTERVENTIONS:
Other: Simulation based curriculum — See arm/group description
  Arms: Simulation based curriculum
Other: Standard training — See arm/group description
  Arms: Standard training

SUMMARY:
TCC-PASTE is a randomised controlled trial comparing a simulation based training curriculum with standard training for ophthalmology residents learning to perform tunnel construction in manual small incision cataract surgery. After obtaining informed consent, participating trainees will be randomly assigned to learn to perform tunnel construction either through the simulation based curriculum or through the standard curriculum at their institute. Trainees assigned to simulation will learn through studying an eBook, participating in training sessions supported by repeated practice on a virtual reality simulator, and supervised training in live surgery to facilitate transfer of skill acquired in simulation to the operating room. To determine the effect of simulation based training, we will assess the number of errors trainees perform in the initial part of their intraoperative learning curve.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a training program at a partner institute;
* No or minimal prior experience with MSICS (trainees within the first 2-3 months of matriculation, or having performed fewer than 20 procedures as the main surgeon but no more than 5 MSICS procedures within 6 months preceding participation in TCC-PASTE);
* Provide informed consent to participate in the study;
* Able to participate in routine patient care activities, as required by the partner institute, without the need to take overnight call for the duration corresponding to the simulation training phase.

Exclusion Criteria:

* Performed scleral tunnel construction as the main surgeon in 20 or more procedures;
* Prior experience with the HelpMeSee simulator or participation in the HelpMeSee simulation training curriculum.
* Required to take overnight call for the duration corresponding to simulation training phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Total surgical errors | 12 weeks
  Incidence of pre-specified errors during tunnel construction through video-based assessment: uveal prolapse (UP), buttonhole incision (BI), premature entry (PE), Descemet's detachment (DD), laceration of upper wall (UL), laceration of lateral walls of tunnel (LL), corneal endothelial touch (ET), contact with iris, (IC) and contact with the lens (LC).

SECONDARY OUTCOMES:
Major surgical errors | 12 weeks
  Incidence of pre-specified errors during tunnel construction through video-based assessment: uveal prolapse (UP), buttonhole incision (BI), premature entry (PE), Descemet's detachment (DD), laceration of upper wall (UL), laceration of lateral walls of tunnel (LL).
Minor surgical errors | 12 weeks
  Incidence of pre-specified errors during tunnel construction through video-based assessment: corneal endothelial touch (ET), contact with iris, (IC) and contact with the lens (LC).
Surgical product/outcome assessment: scleral groove | 12 weeks
  Custom developed structured rating scale; video-based assessment
Surgical product/outcome assessment: tunnel dissection | 12 weeks
  Custom developed structured rating scale; video-based assessment
Surgical product/outcome assessment: paracentesis | 12 weeks
  Custom developed structured rating scale; video-based assessment
Surgical product/outcome assessment: viscoelastic injection/exchange | 12 weeks
  Custom developed structured rating scale; video-based assessment
Surgical product/outcome assessment: keratome entry and extensions | 12 weeks
  Custom developed structured rating scale; video-based assessment
Overall technical skill for tunnel construction | 12 weeks
  Custom developed structured rating scale; video-based assessment
Technical skill: scleral groove | 12 weeks
  Custom developed structured rating scale; video-based assessment
Technical skill: tunnel dissection | 12 weeks
  Custom developed structured rating scale; video-based assessment
Technical skill: paracentesis | 12 weeks
  Custom developed structured rating scale; video-based assessment
Technical skill: viscoelastic injection/exchange | 12 weeks
  Custom developed structured rating scale; video-based assessment
Technical skill: keratome entry and extensions | 12 weeks
  Custom developed structured rating scale; video-based assessment
Task-specific technical skill: scleral tunnel | 12 weeks
  ICO-OSCAR:SICS; video-based assessment
Task-specific technical skill: corneal entry | 12 weeks
  ICO-OSCAR:SICS; video-based assessment
Task-specific technical skill: paracentesis & viscoelastic exchange | 12 weeks
  ICO-OSCAR:SICS; video-based assessment
Global technical skill | 12 weeks
  Global indices in ICO-OSCAR:SICS; video-based assessment

OTHER OUTCOMES:
Incidence of any surgical error or self-reported intervention by supervising surgeon to prevent error | 12 weeks
  Any physical intervention or assistance by supervising surgeon is counted as an additional error
Incidence of major surgical error or self-reported intervention by supervising surgeon to prevent error | 12 weeks
  Any physical intervention or assistance by supervising surgeon is counted as an additional error
Incidence of minor surgical error or self-reported intervention by supervising surgeon to prevent error | 12 weeks
  Any physical intervention or assistance by supervising surgeon is counted as an additional error
Incidence of any physical intervention or assistance by supervising surgeon | 12 weeks
  Each instance of physical intervention or assistance by supervising surgeon is counted as one event.
Incidence of complete intervention or assistance by supervising surgeon | 12 weeks
  Each instance of ake-over by supervising surgeon for the specific activity or rest of task is counted as one event.

CONTACTS AND LOCATIONS:
Locations (1):
- HelpMeSee Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No